CLINICAL TRIAL: NCT03267082
Title: Evaluation the Role of Laparoscopic Management of Perforated Appendicitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, samir hosny mahmoud mohamed, general surgery, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERLMPA
Record Dates: First submitted 2017-08-20; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Perforated Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation the role of Laparoscopic management of perforated a (Experimental)
  Interventions: Other: Laparoscopic management of perforated appendicitis

INTERVENTIONS:
Other: Laparoscopic management of perforated appendicitis — 1. Insertion of Ports
  2. Exposure of the Appendix
  3. peritoneal toilet and aspiration of pus after abdominal exposure
  4. Isolation of Mesoappendicular Artery
  5. Clipping and Dividing of the Artery
  6. Application of 3 x Endoloops
  7. Division of the Appendix
  8. Retrieval of the Appendix in an Endobag

SUMMARY:
A laparoscopic appendectomy (LA) was first reported by Semm in 1983. Since then, its advantages, such as the aesthetic appearance of the wound, less postoperative pain, and faster recovery which facilitates early discharge, have been highlighted, and the number of procedures performed has been continuously increasing.

DETAILED DESCRIPTION:
The LA was performed mostly on uncomplicated appendicitis due to negative opinions about its safety when it was first introduced. However, the application of the procedure has been extended to complicated appendicitis (CA), and it is now considered as an alternative procedure to an open appendectomy (OA) as its safety record has improved . Nevertheless, it is still controversial because there are still concerns about surgical difficulties in managing CA with laparoscopy, overall surgery time, possible post-op complications and conversion to an OA during the surgery.

this study aimed to evaluate the safety and the efficacy of LA for managing perforated appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute perforated appendicitis
* fit for laparoscopy and general anesthesia.
* written informed consent.
* short term outcome data and agree to provide contact information.

Exclusion Criteria:

* high risk for general anesthesia.
* Appendicular abscess and appendicular mass .
* ongoing infections including chest infections .
* Children and pregnant females .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
early recovery | 2 day
  recovery within 2 days

SECONDARY OUTCOMES:
wound cosmetic appearance | 6 months
  no scare of incision post laporscopic mangement

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Semm K. Endoscopic appendectomy. Endoscopy. 1983 Mar;15(2):59-64. doi: 10.1055/s-2007-1021466. PMID 6221925
- [Result] Frazee RC, Bohannon WT. Laparoscopic appendectomy for complicated appendicitis. Arch Surg. 1996 May;131(5):509-11; discussion 511-3. doi: 10.1001/archsurg.1996.01430170055010. PMID 8624197